CLINICAL TRIAL: NCT02179944
Title: Human Chorionic Gonadotropin (hCG) Trend After Medication Abortion: A Prospective Physiologic Study
Brief Title: Human Chorionic Gonadotropin (hCG) Trend After Medication Abortion
Status: Completed | Type: Observational
Sponsor: Planned Parenthood League of Massachusetts (Other)
Responsible Party: Sponsor
Other Study IDs: 2014p000824; SFPRF14-20 (Other Grant/Funding Number: Society for Family Planning Research Fund)
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Undesired Pregnancy
Keywords: medication abortion; serum hCG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants

SUMMARY:
This project will be a prospective physiologic study. We will closely follow 60 medication abortion patients with serial repeat serum hCG and urine semi-quantitative hCG testing. We plan to recruit patients from two gestational age strata: ≤ 49 days and > 49 days.

Study Objectives:

1. To create a nomogram describing the change in serum hCG values in the first five days immediately following medication abortion with mifepristone and misoprostol. Specifically, we will describe the percent serum hCG decline from Day 1 (day of mifepristone) to Day 3 (day after misoprostol), from Day 1 to Day 5, and from Day 1 to Day 7-10.
2. To explore whether there is a significant difference in the rate of hCG decline based on initial gestational age determined by ultrasound and initial serum hCG.
3. To describe the correlation between semi-quantitative urine hCG test results and serum hCG values to determine how soon after initiating medication abortion the urine test can detect completed abortion.

We hypothesize that among successful medication abortions, there will be a predictable trend with at least a 50% drop by Day 3 and 80% drop by Day 5.

ELIGIBILITY:
Inclusion Criteria:

* Desire for medication abortion for pregnancy termination AND
* Pregnancy confirmed by ultrasound and gestational age ≤ 63 days based on transvaginal ultrasound (TVUS) OR
* Positive high-sensitivity urine hCG and intrauterine pregnancy (IUP) not confirmed on TVUS

Exclusion Criteria:

* Ineligibility for medication abortion at Planned Parenthood League of Massachusetts (PPLM) based on current PPLM clinical guidelines
* Initiation of medication abortion on Wednesday or Friday
* Failed pregnancy defined as:

  * Crown-rump length ≥ 7mm and no heartbeat
  * Mean sac diameter ≥ 25mm and no embryo
* Reasonable clinical suspicion for ectopic or molar pregnancy such as abnormal or concerning ultrasound findings
* Multiple gestation
* Age less than 18 years
* Prior participation in this study
* Anticipated inability to present for scheduled follow-up visits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients seeking medication abortion from an outpatient health center
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percent serum hCG decline from Day 1 to Day 3, from Day 1 to Day 5, and from Day 1 to Day 7-10 | 10 days from misoprostol administration
  blood sample collection for hCG testing on Day 3, Day 5 and Day 7-10 (Day 1 is day of mifepristone administration)

SECONDARY OUTCOMES:
difference in rate of hCG decline based on initial gestational age | 10 days after misoprostol administration
  blood sample collection for hCG testing on Day 3, Day 5 and Day 7-10 (Day 1 is day of mifepristone administration)

OTHER OUTCOMES:
how soon after initiating medication abortion a semi-quantitative urine pregnancy test can detect completed abortion | 10 days
  urine sample collection for hCG testing using semi-quantitative urine pregnancy test on Day 1, Day 3, Day 5 and Day 7-10 (Day 1 is day of mifepristone administration)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, MPH, Principal Investigator — PPLM
Locations (1):
- Planned Parenthood, Boston, Massachusetts, United States